CLINICAL TRIAL: NCT05394415
Title: Chemoradiation Plus tisLelizumAb for Conversion Therapy of Locally Nonresectable ESCC
Acronym: LATE
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu Cancer Institute & Hospital (Other)
Responsible Party: Principal Investigator, Hongliang Yu, Dr., Jiangsu Cancer Institute & Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-020-01
Record Dates: First submitted 2022-05-24; First posted 2022-05-27 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Esophageal Squamous Cell Carcinoma; Tislelizumab; Chemoradiation
Keywords: ESCC; Esophageal Squamous Cell Carcinoma; Tislelizumab; Chemoradiation; Conversion therapy; Safty; Efficacy
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — tislelizumab; Paclitaxel; Carboplatin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tislelizumab plus chemoradiation group (Experimental): In the single experimental arm, patients with nonresectable stage IIIb-IVa disease were subjected to receive neoadjuvant tislelizumab (200mg) plus chemoradiation (TP regimen plus 30Gy/12F irradiation) for conversion therapy. If conversion therapy succeeds, patients would proceed to surgery and adjuvant therapy. Otherwise, if patients were still not resectable after the conversion therapy, an additional radiation dose of 15Gy/6F would be scheduled for the ESCC lesions to achieve a definite radiotherapy dose, then, patients proceeded to consolidation therapy.
  Interventions: Drug: Tislelizumab; Drug: Paclitaxel; Drug: Carboplatin; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Tislelizumab — The 1st and 2nd doses were administered concurrently with TP regimen chemotherapy, 200 mg each, on D1 and D22 by intravenous infusion. In patients with successful conversion therapy, one dose of 200 mg on D60, was administered sequentially at the time before surgery after radiation therapy, and two doses of immunotherapy, on D150 and 171, were administered 8 weeks after surgery in concurrent with the 3rd and 4th cycles of chemotherapy as adjuvant therapy; in patients with failed conversion, two doses of chemotherapy combined with tislelizumab, on D60 and D81, were administered 2 weeks after the completion of radiation therapy.
Drug: Paclitaxel — A TP regimen with paclitaxel 135 mg/m^2 + carboplatin AUC=5 was used, on D1 and D22 infused intravenously. Two cycles of adjuvant chemotherapy, on D150, 171, were started 8 weeks after surgery in patients with a successful conversion, and 2 cycles of consolidation chemotherapy, on D60, 81, were started 2 weeks after the end of radiotherapy in patients with unsuccessful conversion therapy.
Drug: Carboplatin — A TP regimen with paclitaxel 135 mg/m^2 + carboplatin AUC=5 was used, on D1, 22 infused intravenously. Two cycles of adjuvant chemotherapy, on D150,171, were started 8 weeks after surgery in patients with a successful conversion, and 2 cycles of consolidation chemotherapy, D60,81, were started 2 weeks after the end of radiotherapy in patients with unsuccessful conversion therapy.
Radiation: Radiotherapy — Radiotherapy was scheduled to be given on D1 of the 2nd cycle of chemotherapy. The primary lesions and/or lymph nodes in the operation area would be radiated in 2 stages. A dose of 30Gy/12F would be given in the first stage. When 12 Fractions were given, our MDT team would evaluate the regression of the lesions according to CT and MR results. If surgery is feasible, radiotherapy would be stopped for the primary lesions and lymph nodes in the operation area; if not resectable, the 2nd stage of radiotherapy would be given with a dose of 15Gy/6F, totaling to 45Gy/18F to the ESCC lesions. Radiotherapy for all lymph nodes outside the operation area was with DT of 45Gy/18F. All radiotherapy in this study was scheduled to be 2.5Gy/F, 1F/d, 5F/w. The preoperative radiotherapy target area was outlined by the consensus of the thoracic surgeon and radiotherapist.

SUMMARY:
This is a single institution and single-arm phase I/II study to assess the feasibility and efficacy of tislelizumab plus chemoradiation for conversion therapy of patients with locally nonresectable ESCC.

DETAILED DESCRIPTION:
The success of PD-1 antibody immunotherapy has brought about tremendous changes in clinical practice for treating patients with ESCC. Many patients with ESCC were not resectable at first presentation because of locally advanced disease in the primary site and/or in lymph nodes. The primary intention of our study was to evaluate the feasibility and efficacy of combining tislelizumab and chemoradiation for conversion therapy for these patients. The enrolled patients in this study should be with pathologically proved ESCC staged IIIb-IVa according to the 8th edition of UICC/AJCC TNM stage classification. This is a single institution and single-arm phase I/II study, the estimated enrollment was 30 participants.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed ESCC；
2. Clinical stage T4 N-/+，or T1-3 N+（IIIb-IVa） (AJCC 8 TNM classiftion);
3. Locally advanced ESCC that are not resectable for primary site and/or lymph nodes evaluated before treatment;
4. At least one measurable lesion in accordance with RECIST 1.1;
5. Have a performance status of 0 or 1 on the ECOG Performance Scale;
6. Expected survival time is greater than 6 months;
7. The important organs' functions meet the following requirements: the absolute neutrophil count(ANC) ≥1.5×10^9/L; the platelet count ≥100×10^9/L; hemoglobin ≥90g/L; bilirubin is less than or equal to 1.5 times ULN, ALT and AST less than or equal 2.5 times UILN; creatinine clearance rate (CCr) ≥50mL/min; the thyroid function is normal;
8. Female subjects of childbearing potential have a negative pregnancy test and must agree to take effective contraceptive measures during the study period and within 3 months after the last dose;
9. Be willing and able to provide written informed consent/assent for the trial.

Exclusion Criteria:

1. The patient has received radiotherapy, chemotherapy, hormone therapy, surgery, or molecular-targeted therapy;
2. Confirmed patients with distant metastasis by CT imaging;
3. The subject has previous or co-existing other malignancies (except cured basal cell carcinoma of the skin and carcinoma in situ of the cervix);
4. The subject had previously received other anti-PD-1 antibody therapy or other immunotherapy targeting PD-1 / PD-L1;
5. Patients with active autoimmune disease or documented autoimmune disease or symptoms requiring systemic hormone therapy or anti-autoimmune drug therapy;
6. Patients with immunodeficiency or who were still receiving systemic steroid hormone therapy (prednisone > 10 mg/ day or other equivalent drugs) or other forms of immunosuppressive therapy 7 days prior to the first dose of neoadjuvant therapy in this study;
7. Clinical ascites or pleural effusion requiring therapeutic puncture or drainage;
8. The subject with uncontrol cardiac clinical symptoms or diseases, such as (1) any class 2 or more heart failure (2) unstable angina pectoris (3) myocardial infarction within 1 year (4) clinically significant ventricular or ventricular arrhythmias requiring treatment or intervention;
9. Abnormal coagulation function (PT>16s, APTT>43s, TT>21s, Fbg> 2G /L), bleeding tendency, or receiving thrombolytic or anticoagulant treatment;
10. The subject is present (within 3 months) with esophageal varices, active gastric and duodenal ulcers, ulcerative colitis, portal hypertension, and other gastrointestinal diseases, or with active bleeding from unresected tumors, or other conditions that may cause gastrointestinal bleeding or perforation as determined by the investigator;
11. Past or present severe bleeding (bleeding >30 ml within 3 months), hemoptysis (fresh blood >5 ml within 4 weeks) or thromboembolism events (including stroke events and/or TRANSIENT ischemic attack) within 12 months;
12. Patients with active infection who still required systemic treatment 7 days before the first dose of neoadjuvant therapy in this study;
13. Patients with past or present objective evidence of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radioactive pneumonia, drug-related pneumonia, severely impaired lung function, etc;
14. Senior or uncontrolled virus injection: HIV, TP, hepatitis virus;
15. Patients who had participated in clinical trials of other drugs within 4 weeks;
16. The live vaccine was administered less than 4 weeks prior to study administration or possibly during the study period;
17. Have a history of mental illness or psychiatric substance abuse;
18. The subject cannot or does not agree to bear the cost of the self-paid portion of the examination and treatment, except for the clinical study drug, combined chemoradiotherapy, and SAE associated with the clinical study drug;
19. Other patients whom the medical practitioner considers inappropriate for inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Treatment safety | up to 2 years
  The incidence and severity of treatment related adverse event according to CTCAE 5.0

SECONDARY OUTCOMES:
Objective response rate (ORR) | up to 2 years
  Objective response rate by assessment per RECIST.
Conversion esophagectomy rate (CER) | up to 2 years
  The ratio of patients succeed to receive esophagectomy after conversion therapy to the number of total patients enrolled in this study and received conversion therapy.
Major pathological response (MPR) | up to 2 years
  Residual viable tumor of less than or equal to 10% in the reseted samples from whom succeed to surgery after the conversion therapy
Progression free survival (PFS) | up to 2 years
  The length of time during and after the enrollment of patients without get worse.
Overall survival (OS) | up to 2 years
  The length of time from the date of enrollment to death for any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Xiangzhi Zhu, Dr., Study Director — Jiangsu Cancer Institute & Hospital
Locations (1):
- Jiangsu Cancer Institute & Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No